CLINICAL TRIAL: NCT01763398
Title: Analysis of the Risk Factors for the Neutropenic Fever in the High Risk NHL Patients for Developing Febrile Neutropenia Who Received 3-weekly CHOP-like Chemotherapy With Primary G-CSF Prophylaxis; Prospective Multicenter Observation Study
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Collaborators: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: 4-2011-0432
Record Dates: First submitted 2013-01-04; First posted 2013-01-08 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- non-Hodgkin's lymphoma: Patients with non-Hodgkin's lymphoma, high risk group for neutropenic fever, treated by CHOP-like regimen and primary G-CSF prophylactic therapy

SUMMARY:
The domestic standards of G-CSF permit the use of the G-CSF only when the ANC(absolute neutrophil count) drops to 1,000/uL or below. Therefore it is impossible to inject the G-CSF in order to prevent neutropenia. However, 'the 2006 Update of Recommendations for the Use of White Blood Cell Growth Factors: An Evidence-Based Clinical Practice Guideline(J ClinOncol 2006; 24:3187-3205)' and the 'NCCN Guideline' have revealed that as a precaution, it is appropriate to inject the G-CSF to the non-Hodgkin's lymphoma patients with high-risk factors under the anticancer treatment of CHOP-21 Rituximab before the number of neutrophils decreases. Thus, it is intended to analyze the risk factors of febrile neutropenia in a high-risk group of non-Hodgkin's lymphoma patients with a neutropenic fever who receive the CHOP-like regimen and primary G-CSF prophylactic therapy every three weeks. (The definition of neutropenic fever is a fever over 38.3 degrees C or continuous fever lasting longer than 1 hour over 38 degrees C with the number of neutrophil ≤ 500/uL or neutrophil ≤ 1,000/uL in case of expected decline to ≤ 500/uL within 48 hours.)

ELIGIBILITY:
Inclusion Criteria:

* Histologically diagnosed non-Hodgkin's lymphoma patients treated by CHOP-regimen or R (Rituximab)-CHOP regimen at 21±5 days interval
* Age >= 20 years old
* The patients with at least one of the following risk factor of neutropenic fever at initiation of anti-cancer treatment

  1. Age >= 65 years old
  2. Progressed stage of disease (Ann Arbor stage III)
  3. History of previous anti-cancer treatment
  4. History of previous radiotherapy (Including bone region includes bone marrow)
  5. Bone marrow involvement
  6. Comorbid neutropenia (neutrophils < 1,500/uL ) before the initiation of anti-cancer treatment
  7. Comorbid anemia (hemoglobin < 12.0 g/dL ) before the initiation of anti-cancer treatment
  8. Evidence of activated inflammation
  9. Existence of open wound
  10. Poor health state (ECOG 2)
  11. Poor nutritional state (Serum albumin < 3.5 g/dL)
  12. Kidney disease or renal insufficiency
  13. Liver disease (chronic hepatitis or cirrhosis) or hepatic insufficiency
  14. Chronic Obstructive Pulmonary Disease (COPD)
  15. Cardiovascular disease
  16. Diabetes mellitus
* Increased cardiac output by 50% above the baseline without clinically significant abnormal findings on MUGA or echocardiography
* life expectancy >=6 months
* Amenorrhea less than 1 year (less than 1 year after menopause) or premenopausal female with negative response to serum or urine pregnancy test before initiation of the treatment
* Voluntary participants with written consent agreement for this study

Exclusion Criteria:

* The patients treated by other anti-cancer treatment except CHOP regimen or R (Rituximab)-CHOP regimen at 21 days interval
* Pregnant or breast feeding woman, fertile woman without appropriate contraception
* Patients with hypersensitivity against study drugs
* Patients treated by other study medication or co-treatment with anticancer chemotherapy, hormone therapy, and immunotherapy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-Hodgkin's lymphoma, high risk group for neutropenic fever, treated by CHOP-like regimen and primary G-CSF prophylactic therapy
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2011-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Hospitalization period | 24months
  Hospitalization relevant to this during the occurrence of febrile neutropenia under anticancer treatments

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, Seoul, South Korea